CLINICAL TRIAL: NCT02548637
Title: Effects of Acupuncture on Aromatase Inhibitor-Induced Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACU-JOINT001
Record Dates: First submitted 2015-06-18; First posted 2015-09-14 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture Therapy (Experimental): Based on the Traditional Chinese Medicine theory, investigators will use the systemic treatment methods (full body treatment with the joint specifications). Every patient will receive the standard protocols of these points uniformly regardless of their symptoms. The only variable will be the location of placement of the four electrodes (two positive charges and two negative charges) to the needle points at the most painful joints bilaterally. Needles will be in place a total of 45 minutes per session. The Thermal Design Power (TDP) infrared heat lamp will be applied concurrently to the most painful joint(s) for the entire 45 minutes. Acupuncture will be administered twice a week for 6 weeks, then once a week for an additional 4 weeks.
  Interventions: Procedure: Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture Therapy — The standard textbook of Chinese Acupuncture and Moxibustion is the source for the name and location of the points for this study. A total of 38 points will be used, divided between two acupuncture sessions: 20 points or 37 locations in the supine position; 18 points or 36 locations in the prone position. Other than points governing vessel (GV) 20, conception vessel (CV) 6, CV 10, all points will be performed bilaterally.

SUMMARY:
Researchers at the John Wayne Cancer Institute (JWCI) at Providence Saint John's Health Center (PSJHC) are trying to examine whether acupuncture reduces joint pain in patients being treated with aromatase inhibitor (AI) therapy for breast cancer and whether the reduction in pain happens by lowering inflammation.

DETAILED DESCRIPTION:
The investigators propose to investigate the effect of acupuncture on patients experiencing joint pain from aromatase inhibitor therapy. The investigators will serially measure patient's symptoms and track current medications, joint pain, daily activities, fatigue, and quality of life. The investigators will collect peripheral blood at baseline, weeks 4 and 7, one week after the last acupuncture treatment and 4 weeks after the last acupuncture treatment. The investigators will study the samples collected at the five predetermined time-points to test for immune parameters, such as the innate and adaptive immune responses, as well as the proliferative capabilities and pro-inflammatory mediators reflected in innate and adaptive functional immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Must be on aromatase inhibitor therapy continuously for breast cancer treatment for at least the preceding two months
* Must have experienced increased or new onset joint pain daily to a degree equal to or greater than 4 on a pain scale of 0-10 after starting aromatase inhibitor therapy
* Able to read and write English
* Able to give written informed consent to participate in the study

Exclusion Criteria:

* Have a known autoimmune disease or acute infection
* Have had acupuncture treatment within 6 months of study enrollment
* Known needle phobia
* Known metal allergies
* Have an implantable device, such as pacemaker, defibrillator or other device contraindicated with electrical stimulation
* Use of nonsteroidal antiinflammatory drugs (NSAIDs) or narcotics within 7 days of study enrollment and during study period (15 weeks)
* Receipt of prior chemotherapy, immunotherapy or radiation therapy within 90 days
* On anticoagulant therapy
* Receiving physical or occupational therapy concurrently
* Taking herbs or herbal teas within 7 days of study enrollment and during study period (15 weeks)
* Have an immune-compromising medical condition or currently receiving immune-modulating therapies (including corticosteroids)
* Enrolled in any other active cancer treatment protocols
* Bone fracture or surgery of an affected extremity within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Joint Pain tabulated from Joint Pain Assessment Questionnaire | 3 years
  Investigators will serially measure joint pain symptoms using questionnaires administered at pre-determined time points. A summary of pain scores will be tabulated for all visits.

SECONDARY OUTCOMES:
Adaptive immune response as measured by cytokine levels | 3 years
  Investigators will collect prospective blood samples to test for for cytokine levels
Innate immune response as measured by cytokime levels | 3 years
  Investigators will collect prospective blood samples to test for cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Crane-Okada, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No